CLINICAL TRIAL: NCT00808158
Title: Metabolic Syndrome in Adolescents: Contribution of Tobacco and Central Fat
Brief Title: Examining the Relationship Between Tobacco Exposure, Abdominal Obesity, and Metabolic Syndrome in Adolescents (The STRONG Kids Study)
Acronym: STRONG Kids
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Stephen Cook, Associate Professor, University of Rochester
Other Study IDs: 612; R01HL083056-01 (NIH); HL086946-02
Record Dates: First submitted 2008-12-12; First posted 2008-12-15 (Estimated); Last update posted 2012-11-30 (Estimated); Status verified 2012-11

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, whole blood, white blood cells, saliva, urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Children ages 9 to 10 years old, with a body mass index (BMI) in the 50th to 98th percentile range

SUMMARY:
Metabolic syndrome is a term that describes a group of conditions that increase the risk of cardiovascular disease. The conditions include high blood pressure, obesity, and high cholesterol. This study will examine how changes in tobacco exposure and weight can affect the risk of developing metabolic syndrome among adolescents.

DETAILED DESCRIPTION:
Metabolic syndrome is a term that is used to describe a group of risk factors for cardiovascular disease. The risk factors include obesity, insulin resistance, high cholesterol, and high blood pressure. Two of the most common risk factors for cardiovascular disease-tobacco exposure and abdominal obesity-are also known to influence the development of metabolic syndrome. Metabolic syndrome risk factors, as well as higher obesity levels, are being observed increasingly in adolescents. It is important to understand the relationship between tobacco exposure, abdominal obesity, and metabolic syndrome during early adolescence, as this time period is when lifestyle habits, including diet, exercise, and tobacco use, develop. The purpose of the study is to determine how changes in abdominal obesity and tobacco exposure among adolescents affect the development of metabolic syndrome risk factors, including glucose intolerance and increased levels of cholesterol and blood pressure.

This 3-year study will enroll children with a body mass index in the 50th to 98th percentile and one of their parents. At a baseline study visit, children and parents will complete questionnaires on health, nutrition, physical activity, smoke exposure, and stress levels. Children will undergo a blood and saliva collection; physical examination; measurements of blood pressure, height, weight, and waist circumference; a dual-energy x-ray absorptiometry (DEXA) scan to measure body fat and muscle; and skin fold measurements to measure body fat. Parents will undergo a saliva collection and measurements of blood pressure, height, weight, and waist circumference. Some children will wear an activity monitor for 7 days, and some children will complete a glucose tolerance test, which will involve an additional blood collection. Every 6 months, study researchers will contact parents to confirm the family's contact information. Once a year for 3 years, all participants will complete questionnaires and a saliva collection. Additionally, at Year 3, all participants will also undergo repeat measurements of blood pressure, height, weight, and waist circumference.

ELIGIBILITY:
Inclusion Criteria:

* BMI in the 50th to 98th percentile range
* Parent or caregiver must agree to participate in the study

Exclusion Criteria for All Participants:

* Inability to speak and understand English
* Family residence outside the greater Rochester area (more than 50 miles from the clinical research center)
* Family is planning to leave the greater Rochester area (move more than 50 miles from the clinical research center) in the 24 months after study entry

Exclusion Criteria for Children:

* Significant medical condition, including cystic fibrosis, type 1 or type 2 diabetes, or other conditions that could interfere with the assessment of metabolic-related outcome measures
* Tanner stage 3 or greater
* Currently taking medications that alter appetite and/or glucose metabolism

Ages: 9 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: A community sample of 240 9- to 10-year olds with varying abdominal obesity levels (all having a waist circumference equal to or above the 50th percentile for age and gender) and varying tobacco smoke exposure levels (from none to high levels)
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2008-10; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Baseline association between tobacco exposure, abdominal obesity, adiponectin, and metabolic syndrome components | Measured at baseline

SECONDARY OUTCOMES:
Temporal change in abdominal obesity, adiponectin, and metabolic syndrome components, as correlated with level of tobacco exposure | Measured at Years 1, 2, and 3

CONTACTS AND LOCATIONS:
Overall Officials: Stephen R. Cook, MD, MPH, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States